CLINICAL TRIAL: NCT02413229
Title: A Randomized Double Blind Vehicle Controlled Dose Ranging Multiple Site Phase 2 Clinical Study to Evaluate the Efficacy and Safety of DSXS in Patients With Moderate to Severe Scalp Psoriasis
Brief Title: A Randomized Double Blind Vehicle Controlled Dose Ranging Parallel Design Multiple Site Clinical Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSXS 1411
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DSXS1411 (Experimental): DSXS applied once a day for a total of 28 days.
  Interventions: Drug: DSXS1411
- Placebo (Placebo Comparator): Placebo (vehicle) applied once a day for a total of 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DSXS1411 — DSXS (Taro Pharmaceuticals Inc.)
  Other Names: Active
  Arms: DSXS1411
Drug: Placebo — Placebo (vehicle) (Taro Pharmaceuticals Inc.)
  Other Names: vehicle
  Arms: Placebo

SUMMARY:
The objectives of this study are to evaluate the therapeutic efficacy and safety of DSXS and a Placebo in patients with moderate to severe scalp psoriasis.

DETAILED DESCRIPTION:
This randomized, double-blind, vehicle-controlled, dose-ranging, parallel-group multi-site study is designed to evaluate the therapeutic efficacy and safety of the investigational product, DSXS, for the treatment of moderate to severe scalp psoriasis at different application times up to 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females age 12 and older.
* Clinical diagnosis of moderate to severe scalp psoriasis, defined by a Investigator's Global Assessment score of at least 3 at screening.

Exclusion Criteria:

* Under 12 years of age.
* Patients whose scalp and/or non-scalp psoriasis necessitates systemic or other concomitant topical therapies during the study.
* Has a scalp skin condition that would interfere with the diagnosis or assessment of plaque psoriasis of the scalp.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-09-14 (Actual); Study Completion 2016-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novum Pharmaceutical Research Services, Study Chair — http://www.novumprs.com/contact

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DSXS1411 5 Min: DSXS applied once a day for a total of 28 days for duration of 5 minutes.
  DSXS1411: DSXS (Taro Pharmaceuticals Inc.)
- Placebo 5 Min: Placebo (vehicle) applied once a day for a total of 28 days for duration of 5 minutes.
  Placebo: Placebo (vehicle) (Taro Pharmaceuticals Inc.)
- DSXS1411 10 Min: DSXS applied once a day for a total of 28 days for duration of 10 minutes.
  DSXS1411: DSXS (Taro Pharmaceuticals Inc.)
- Placebo 10 Min: Placebo (vehicle) applied once a day for a total of 28 days for duration of 10 minutes.
  Placebo: Placebo (vehicle) (Taro Pharmaceuticals Inc.)
- DSXS1411 15 Min: DSXS applied once a day for a total of 28 days for duration of 15 minutes.
  DSXS1411: DSXS (Taro Pharmaceuticals Inc.)
- Placebo 15 Min: Placebo (vehicle) applied once a day for a total of 28 days for duration of 15 minutes.
  Placebo: Placebo (vehicle) (Taro Pharmaceuticals Inc.)
- DSXS1411 30 Min: DSXS applied once a day for a total of 28 days for duration of 30 minutes.
  DSXS1411: DSXS (Taro Pharmaceuticals Inc.)
- Placebo 30 Min: Placebo (vehicle) applied once a day for a total of 28 days for duration of 30 minutes.
  Placebo: Placebo (vehicle) (Taro Pharmaceuticals Inc.)
Period: Overall Study
Arm/Group | DSXS1411 5 Min | Placebo 5 Min | DSXS1411 10 Min | Placebo 10 Min | DSXS1411 15 Min | Placebo 15 Min | DSXS1411 30 Min | Placebo 30 Min
Started | 25 | 12 | 26 | 12 | 24 | 12 | 25 | 15
Completed | 24 | 11 | 25 | 11 | 21 | 12 | 25 | 11
Not Completed | 1 | 1 | 1 | 1 | 3 | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DSXS1411 5 Min | Placebo 5 Min | DSXS1411 10 Min | Placebo 10 Min | DSXS1411 15 Min | Placebo 15 Min | DSXS1411 30 Min | Placebo 30 Min | Total
Number analyzed (Participants) | 24 | 12 | 26 | 12 | 22 | 12 | 25 | 15 | 148
Age, Customized [Count of Participants; unit: Participants]
  < 18 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 5
  18 - 40 | 6 | 4 | 5 | 5 | 4 | 6 | 5 | 10 | 45
  41 - 64 | 13 | 4 | 18 | 5 | 14 | 5 | 13 | 4 | 76
  65 - 75 | 3 | 3 | 3 | 0 | 4 | 1 | 4 | 1 | 19
  > 75 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 19 | 7 | 14 | 8 | 12 | 10 | 92
  Male | 12 | 2 | 7 | 5 | 8 | 4 | 13 | 5 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 4 | 8 | 4 | 7 | 5 | 7 | 4 | 48
  Not Hispanic or Latino | 15 | 8 | 18 | 8 | 15 | 7 | 18 | 11 | 100
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 2 | 0 | 0 | 1 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3
  White | 23 | 10 | 24 | 9 | 22 | 11 | 23 | 15 | 137
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Time Patient has Suffered from Symptoms [Count of Participants; unit: Participants]
  < 3 Months | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  3 to 6 Months | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  6 to 12 Months | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 2 | 10
  > 1 Year And <= 3 Years | 3 | 3 | 3 | 4 | 6 | 4 | 3 | 3 | 29
  > 3 Years And <= 5 Years | 4 | 0 | 6 | 1 | 3 | 1 | 2 | 4 | 21
  > 5 Years | 13 | 8 | 16 | 4 | 12 | 6 | 19 | 5 | 83

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response of Success
Description: The proportion of patients in each treatment group that have clinical success at Day 28, which is defined by a Investigator's Global Assessment score of 0 or 1.
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS1411 5 Min | Placebo 5 Min | DSXS1411 10 Min | Placebo 10 Min | DSXS1411 15 Min | Placebo 15 Min | DSXS1411 30 Min | Placebo 30 Min
Number analyzed (Participants) | 24 | 12 | 26 | 12 | 22 | 12 | 25 | 15
Participants | 6 | 4 | 6 | 1 | 6 | 1 | 11 | 1
Statistical Analysis 1: Comparison: DSXS1411 5 Min vs Placebo 5 Min; Test type: Superiority; p = 0.3571, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: DSXS1411 10 Min vs Placebo 10 Min; Test type: Superiority; p = 0.5224, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: DSXS1411 15 Min vs Placebo 15 Min; Test type: Superiority; p = 0.3890, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: DSXS1411 30 Min vs Placebo 30 Min; Test type: Superiority; p = .0325, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | DSXS1411 5 Min | Placebo 5 Min | DSXS1411 10 Min | Placebo 10 Min | DSXS1411 15 Min | Placebo 15 Min | DSXS1411 30 Min | Placebo 30 Min
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/12 | 0/26 | 0/12 | 0/22 | 0/12 | 0/25 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/12 | 0/26 | 0/12 | 0/22 | 0/12 | 0/25 | 0/15
Other Adverse Events (participants affected / at risk) | 4/24 | 3/12 | 3/26 | 3/12 | 4/22 | 4/12 | 7/25 | 5/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DSXS1411 5 Min (N=24) | Placebo 5 Min (N=12) | DSXS1411 10 Min (N=26) | Placebo 10 Min (N=12) | DSXS1411 15 Min (N=22) | Placebo 15 Min (N=12) | DSXS1411 30 Min (N=25) | Placebo 30 Min (N=15)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Application site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Application site pruritis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear swelling (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Hepatic enzyme increased (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes